CLINICAL TRIAL: NCT03888079
Title: Patient Satisfaction After Surgery for Otosclerosis Under Local ou General Anesthesia
Acronym: SPOC
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3061_SPOC
Record Dates: First submitted 2019-02-04; First posted 2019-03-25 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2019-03

CONDITIONS: Otosclerosis; Otosclerosis Surgery
Keywords: Otosclerosis; otosclerosis surgery; local anesthesia; general anesthesia; comfort assessment; Glasgow Benefit Inventory questionnaire; hearing results
MeSH Terms: conditions — Otosclerosis | interventions — Anesthetics, Local; Anesthetics, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Local anesthetic: Patients who chose local anesthesia for their surgery
  Interventions: Drug: Local anesthetic
- General anesthetic: Patients who chose general anesthesia for their surgery
  Interventions: Drug: general anesthetic

INTERVENTIONS:
Drug: Local anesthetic — 1% or 2% lidocaine with 1:100,000 epinephrine, augmented by intravenous sedation and analgesia
  Groups: Local anesthetic
Drug: general anesthetic — Endotracheal intubation, intravenous narcotic agents, and inhaled agents
  Groups: General anesthetic

SUMMARY:
Main purpose of this study is to compare comfort level of patients, after otosclerosis surgery, under local or general anesthesia.

DETAILED DESCRIPTION:
The care system will not differ from the usually treatment of patients. Patients will decided about the type of anesthesia (local or general) after detailed description of both procedures.

All operations will be performed by the same surgeon and the same basic surgical technique.

The only difference is that patients included in thi study will have to complete a satisfactory survey 10 days after surgery and a GBI questionnaire 3 months after surgery, during the post operative consultations .

ELIGIBILITY:
Inclusion criteria:

* Patients older than 18 years suffering from otosclerosis who have surgical indication.
* Patients who want surgical treatment for their otosclerosis
* Clinic : Deafness with social prejudice and normal otoscopic exam
* Audiometric : conductive or mixed hearing loss with abolition of the aural reflex. Audiometric threshold more than 30decibel (dB) and air bone gap more important than 20dB.
* Pré operative scan in favor of otosclerosis
* Diagnosis confirmation during the surgery with stapes sclerotic's attachments to the oval window

Exclusion criteria:

* History of ear surgery
* No medical objection to local anesthesia
* No medical objection to general anesthesia
* No medical objection to ear surgery
* No legal protection for adults
* No participation refusal

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from otosclerosis who have surgical indication
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Visual comfort scale (EVA type ruler) | 10 days after surgery
  respondents specify their level of comfort during the surgery by indicating a position along a continuous line between two end-points : Minimum score is 0 (no comfort) and maximum is 10 (very comfortable) during surgery

SECONDARY OUTCOMES:
Glasgow Benefit Inventory questionnaire GBI | 3 months after surgery
  Glasgow Benefit Inventory questionnaire GBI (GBI, Robinson et al. 1996).
  * The Glasgow Benefit Inventory (GBI) is a measure of patient benefit developed especially for otorhinolaryngological (ORL) interventions.
    18 items in 3 categories defined by social, psychological, and physical perceptions of well-being
  * Responses are based on a 5-point Likert scale, ranging from a large deterioration in health status (1) to a large improvement (5).
  * The total GBI score is then calculated from an average of the Likert scores to give equal weight to each question. The average (1 5) is subtracted by 3 (no change), and the result is multiplied by 50 to produce a GBI score that ranges from 100 (maximum detriment after surgery) to 100 (maximum improvement after the intervention). A GBI score of zero is neutral and indicates no improvement or detriment from the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Godey, PH-PD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France